CLINICAL TRIAL: NCT01646853
Title: Radiation Dose Study of Concurrent Chemoradiotherapy With Cisplatin Plus Fluorouracil in Oesophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: JSNT0415
Record Dates: First submitted 2012-07-09; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms

ARMS (1):
- Concurrent radiochemotherapy (Experimental)
  Interventions: Radiation: Megavoltage photon beam; Drug: cisplatin-fluorouracil chemotherapy

INTERVENTIONS:
Radiation: Megavoltage photon beam — initial dose:50Gy/2Gy/25f,5days/week escalation dose:4Gy/2Gy/2f
Drug: cisplatin-fluorouracil chemotherapy — cisplatin 75 mg/m2 on day 1 with standard hydration fluorouracil 1000 mg/m2/day1 i.v. by continuous infusion from day 1 to day 4 of each cycle
  Other Names: PF chemotherapy

SUMMARY:
The objective of this study is to determine the optimal radiation dosage used in concurrent chemo-radiotherapy in Chinese population. A dose climbing experiment is carried out with an initiate dose of 50Gy conventionally applied in Western countries.

DETAILED DESCRIPTION:
Esophageal cancer (EC) continues to be a major health burden worldwide. The 5-year survival rates for esophageal cancer have remained less than 15% over decades, probably because of ineffective therapies and the detection of late-stage cancers. Concurrent chemo-radiotherapy was established as one of the viable options for therapy of patients with localized EC following the results from the landmark trial of the Radiation Therapy Oncology Group (RTOG) 85-01 trial, showing a significant survival advantage of concurrent chemoradiation over radiation alone.

The use of radiochemotherapy with cisplatin and 5-fluorouracil (5-FU) is a well-accepted standard for the definitive treatment of esophageal cancer in China which has also been demonstrated efficacy and good tolerability internationally. The AJCC recommended dose range of radiotherapy for concurrent therapy is 45-50.4Gy. Moreover, (RTOG) 85-01 trial also established 50.4 Gy as the standard dose of radiation to be administered concurrently with chemotherapy. However, the appropriate dose of radiation fit for Chinese remains controversial. Due to insufficient evidence of EBM, radiation therapist in China always prescribe a radiation dosage by their own experience. Dosages (e.g. 60-64Gy) significantly higher than the international standard is commonly used in Chinese EC patients which lead to a greater likelihood of toxicity. Thus Chinese oncologists are urgent to reach a consensus about radiation dosage in the standard treatment of local advanced EC.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven squamous cell carcinoma or adenocarcinoma of thoracic or cervical esophagus or gastroesophageal junction esophagus, including the gastroesophageal junction
2. Measurable lesion
3. Age > 18 years
4. Karnofsky performance score > 70
5. Life expectancy > 3 months
6. Adequate bone marrow function (white blood cell [WBC] count ≥ 3.5 109/L, neutrophil count ≥ 2.0 109/L, and platelet count ≥ 100 109/L), adequate renal function (creatinine ≤ 2 mg/dL or creatinine clearance ≥ 50 mL/min), and normal liver function (aspartate aminotransferase and alanine aminotransferase less than two times the upper limit of normal, total serum bilirubin ≤ 1.5 mg/dL).

Exclusion Criteria:

1. Prior systemic chemotherapy for EC
2. Evidence of distant metastatic disease
3. Evidence of uncontrolled medical conditions (e.g.,serious infection,grade 4 hypertension,congestive heart failure)
4. A history of concomitant or previous malignancy.
5. Physical evidence of peripheral neuropathy or hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor Response | One day after completion of the initial therapeutic dose (50.0Gy) and the total dose of radiotherapy
  objective evaluation is made according to the standards of Response Evaluation Criteria in Solid Tumors (RECIST)，defined as complete response(CR),partial response (PR)，stable disease(SD),and progressive disease (PD).Tumor sizes are measured using barium esophagram or CT.

SECONDARY OUTCOMES:
adverse events | Side effect assessment was performed every week for the duration of concurrent radiochemotherapy, an expected average of 5 weeks
  using the National Cancer Institute Common Toxicity Criteria,predominantly observe the presence of radiation esophagitis,radiaion pneumonia and hematological toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Xinchen Sun, M.D.,Ph.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China